CLINICAL TRIAL: NCT04266457
Title: Establishing Alpha-synuclein Real Time - Quaking Induced Conversion (RT-QuIC) Assay as a Diagnostic Technique in Rapid Eye Movement (REM) Sleep Behaviour Disorder (RBD)
Brief Title: Establishing Alpha-synuclein RT-QuIC Assay as a Diagnostic Technique in REM Sleep Behaviour Disorder
Status: Withdrawn | Type: Observational
Why Stopped: Study stopped after ethical approval but before first patient gave consent due to pandemic
Sponsor: University of Edinburgh (Other)
Collaborators: Weston Brain Institute (Other)
Responsible Party: Sponsor
Other Study IDs: AC20015
Record Dates: First submitted 2020-02-10; First posted 2020-02-12 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2021-05

CONDITIONS: Sleep Disorder Rem Sleep Behavior; Parkinson's Disease, Lewy Body
Keywords: REMBD; REM Behavioural Disorder; prodromal α-synucleinopathies
MeSH Terms: conditions — REM Sleep Behavior Disorder; Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — 5ml ceberospinal fluid, 9ml blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No Intervention — No Intervention

SUMMARY:
We hypothesise that a real-time quaking induced conversion assay for the detection of pathological alpha-synuclein (α -syn RTQuIC) can be used to differentiate between cases of idiopathic REM-sleep behaviour disorder (RBD) and RBD that is symptomatic of prodromal α-synucleinopathies.

DETAILED DESCRIPTION:
This study will be the largest analysis of cerebrospinal fluid (CSF) α-synuclein in Rapid Eye Movement Behaviour Disorder (RBD) patients to date. In line with the The National CJD Research & Surveillance Unit (NCJDRSU)'s recent inclusion of a positive RT-QuIC for pathological prion protein in the diagnostic criteria for Creutzfeldt-Jakob Disease (CJD) [1], we aim to deploy this novel method to establish it as an accurate research and diagnostic resource in the assessment and prognosis of RBD. This research is transformative and has the potential to change practice.

Currently, there is no simple method with high sensitivity and specificity available which can identify patients who will go on to develop an α - synucleinopathy. Clinical assessment of a panel of markers (e.g. Postuma et al. 2015) are time-consuming and impractical in normal clinical settings, with the majority of patients presenting to sleep physicians, geriatricians, and non-specialised neurology clinics, both publicly and privately. This has a major impact on counselling strategies for RBD patients, appropriate follow-up, trials of novel neuro-protective agents in alpha-synucleinopathies before full-blown phenotype is manifest and enhancing understanding of pathways involved in RBD out-with the dopaminergic system.

RBD is a common, sometimes fatal disease (through injury to self/others) and treatments are indiscriminate regarding aetiology with limited evidence-base. A simple test using CSF (analogous to measuring CSF-orexin levels to diagnose narcolepsy+cataplexy) with high sensitivity and specificity is ideal. Thus, we believe that the central thesis of our work will not only inform subsequent behavioural, genetic and neuroimaging characterisation of our established RBD cohort, but will also translate the α-syn RT-QuIC concept into evidence-based and effective clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Rapid Eye Movement Behaviour Disorder (RBD) using the International Classification of Sleep Disorders version 3 (ICSD-3) criteria [18] - Patients aged 18 years and over - Patient able to give written informed consent

Exclusion Criteria:

* RBD secondary to medication or withdrawal state. - <18 years old - Inability to give written informed consent - Contraindication to lumbar puncture procedure (e.g. patients taking Warfarin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with REM Sleep Behavioural Disorder using ICSD-3 criteria
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Presence of pathological α-synuclein within the cerebrospinal fluid (CSF) | 0-24 months after sample taken
  The primary outcome measure will be either a positive/negative (binary) result from the α-syn RT-QuIC assay. A positive output confirms presence of pathological α-synuclein within the CSF.

CONTACTS AND LOCATIONS:
Overall Officials: Renata L Riha, MD, Principal Investigator — University of Edinburgh
Locations (1):
- The University of Edinburgh, Edinburgh, Lothian, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Postuma RB, Gagnon JF, Bertrand JA, Genier Marchand D, Montplaisir JY. Parkinson risk in idiopathic REM sleep behavior disorder: preparing for neuroprotective trials. Neurology. 2015 Mar 17;84(11):1104-13. doi: 10.1212/WNL.0000000000001364. Epub 2015 Feb 13. PMID 25681454
- [Background] Iranzo A, Tolosa E, Gelpi E, Molinuevo JL, Valldeoriola F, Serradell M, Sanchez-Valle R, Vilaseca I, Lomena F, Vilas D, Llado A, Gaig C, Santamaria J. Neurodegenerative disease status and post-mortem pathology in idiopathic rapid-eye-movement sleep behaviour disorder: an observational cohort study. Lancet Neurol. 2013 May;12(5):443-53. doi: 10.1016/S1474-4422(13)70056-5. Epub 2013 Apr 3. PMID 23562390
- [Background] Boeve BF, Silber MH, Ferman TJ, Lin SC, Benarroch EE, Schmeichel AM, Ahlskog JE, Caselli RJ, Jacobson S, Sabbagh M, Adler C, Woodruff B, Beach TG, Iranzo A, Gelpi E, Santamaria J, Tolosa E, Singer C, Mash DC, Luca C, Arnulf I, Duyckaerts C, Schenck CH, Mahowald MW, Dauvilliers Y, Graff-Radford NR, Wszolek ZK, Parisi JE, Dugger B, Murray ME, Dickson DW. Clinicopathologic correlations in 172 cases of rapid eye movement sleep behavior disorder with or without a coexisting neurologic disorder. Sleep Med. 2013 Aug;14(8):754-62. doi: 10.1016/j.sleep.2012.10.015. Epub 2013 Mar 7. PMID 23474058
- [Background] Schenck CH, Boeve BF, Mahowald MW. Delayed emergence of a parkinsonian disorder or dementia in 81% of older men initially diagnosed with idiopathic rapid eye movement sleep behavior disorder: a 16-year update on a previously reported series. Sleep Med. 2013 Aug;14(8):744-8. doi: 10.1016/j.sleep.2012.10.009. Epub 2013 Jan 22. PMID 23347909
- [Background] Plomhause L, Dujardin K, Duhamel A, Delliaux M, Derambure P, Defebvre L, Monaca Charley C. Rapid eye movement sleep behavior disorder in treatment-naive Parkinson disease patients. Sleep Med. 2013 Oct;14(10):1035-7. doi: 10.1016/j.sleep.2013.04.018. Epub 2013 Jul 25. PMID 23890957
- [Background] Braak H, Del Tredici K, Rub U, de Vos RA, Jansen Steur EN, Braak E. Staging of brain pathology related to sporadic Parkinson's disease. Neurobiol Aging. 2003 Mar-Apr;24(2):197-211. doi: 10.1016/s0197-4580(02)00065-9. PMID 12498954
- [Background] Kim YK, Yoon IY, Kim JM, Jeong SH, Kim KW, Shin YK, Kim BS, Kim SE. The implication of nigrostriatal dopaminergic degeneration in the pathogenesis of REM sleep behavior disorder. Eur J Neurol. 2010 Mar;17(3):487-92. doi: 10.1111/j.1468-1331.2009.02854.x. Epub 2009 Nov 24. PMID 19968708
- [Background] Barber TR, Lawton M, Rolinski M, Evetts S, Baig F, Ruffmann C, Gornall A, Klein JC, Lo C, Dennis G, Bandmann O, Quinnell T, Zaiwalla Z, Ben-Shlomo Y, Hu MTM. Prodromal Parkinsonism and Neurodegenerative Risk Stratification in REM Sleep Behavior Disorder. Sleep. 2017 Aug 1;40(8):zsx071. doi: 10.1093/sleep/zsx071. PMID 28472425
- [Background] Puschmann A, Bhidayasiri R, Weiner WJ. Synucleinopathies from bench to bedside. Parkinsonism Relat Disord. 2012 Jan;18 Suppl 1:S24-7. doi: 10.1016/S1353-8020(11)70010-4. PMID 22166445
- [Background] Peelaerts W, Baekelandt V. a-Synuclein strains and the variable pathologies of synucleinopathies. J Neurochem. 2016 Oct;139 Suppl 1:256-274. doi: 10.1111/jnc.13595. Epub 2016 Mar 30. PMID 26924014
- [Background] Tyson T, Steiner JA, Brundin P. Sorting out release, uptake and processing of alpha-synuclein during prion-like spread of pathology. J Neurochem. 2016 Oct;139 Suppl 1(Suppl 1):275-289. doi: 10.1111/jnc.13449. Epub 2016 Feb 10. PMID 26617280
- [Background] El-Agnaf OM, Salem SA, Paleologou KE, Curran MD, Gibson MJ, Court JA, Schlossmacher MG, Allsop D. Detection of oligomeric forms of alpha-synuclein protein in human plasma as a potential biomarker for Parkinson's disease. FASEB J. 2006 Mar;20(3):419-25. doi: 10.1096/fj.03-1449com. PMID 16507759
- [Background] Tinsley RB, Kotschet K, Modesto D, Ng H, Wang Y, Nagley P, Shaw G, Horne MK. Sensitive and specific detection of alpha-synuclein in human plasma. J Neurosci Res. 2010 Sep;88(12):2693-700. doi: 10.1002/jnr.22417. PMID 20648655
- [Background] Foulds PG, Mitchell JD, Parker A, Turner R, Green G, Diggle P, Hasegawa M, Taylor M, Mann D, Allsop D. Phosphorylated alpha-synuclein can be detected in blood plasma and is potentially a useful biomarker for Parkinson's disease. FASEB J. 2011 Dec;25(12):4127-37. doi: 10.1096/fj.10-179192. Epub 2011 Aug 24. PMID 21865317
- [Background] Doppler K, Jentschke HM, Schulmeyer L, Vadasz D, Janzen A, Luster M, Hoffken H, Mayer G, Brumberg J, Booij J, Musacchio T, Klebe S, Sittig-Wiegand E, Volkmann J, Sommer C, Oertel WH. Dermal phospho-alpha-synuclein deposits confirm REM sleep behaviour disorder as prodromal Parkinson's disease. Acta Neuropathol. 2017 Apr;133(4):535-545. doi: 10.1007/s00401-017-1684-z. Epub 2017 Feb 8. PMID 28180961
- [Background] Fairfoul G, McGuire LI, Pal S, Ironside JW, Neumann J, Christie S, Joachim C, Esiri M, Evetts SG, Rolinski M, Baig F, Ruffmann C, Wade-Martins R, Hu MT, Parkkinen L, Green AJ. Alpha-synuclein RT-QuIC in the CSF of patients with alpha-synucleinopathies. Ann Clin Transl Neurol. 2016 Aug 28;3(10):812-818. doi: 10.1002/acn3.338. eCollection 2016 Oct. PMID 27752516
- [Background] Li SX, Wing YK, Lam SP, Zhang J, Yu MW, Ho CK, Tsoh J, Mok V. Validation of a new REM sleep behavior disorder questionnaire (RBDQ-HK). Sleep Med. 2010 Jan;11(1):43-8. doi: 10.1016/j.sleep.2009.06.008. Epub 2009 Nov 30. PMID 19945912
- [Background] Johns MW. A new method for measuring daytime sleepiness: the Epworth sleepiness scale. Sleep. 1991 Dec;14(6):540-5. doi: 10.1093/sleep/14.6.540. PMID 1798888
- [Background] Holmes TH, Rahe RH. The Social Readjustment Rating Scale. J Psychosom Res. 1967 Aug;11(2):213-8. doi: 10.1016/0022-3999(67)90010-4. No abstract available. PMID 6059863
- [Background] Goetz CG, Tilley BC, Shaftman SR, Stebbins GT, Fahn S, Martinez-Martin P, Poewe W, Sampaio C, Stern MB, Dodel R, Dubois B, Holloway R, Jankovic J, Kulisevsky J, Lang AE, Lees A, Leurgans S, LeWitt PA, Nyenhuis D, Olanow CW, Rascol O, Schrag A, Teresi JA, van Hilten JJ, LaPelle N; Movement Disorder Society UPDRS Revision Task Force. Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS): scale presentation and clinimetric testing results. Mov Disord. 2008 Nov 15;23(15):2129-70. doi: 10.1002/mds.22340. PMID 19025984
- [Background] White C, Hill EA, Morrison I, Riha RL. Diagnostic delay in REM sleep behavior disorder (RBD). J Clin Sleep Med. 2012 Apr 15;8(2):133-6. doi: 10.5664/jcsm.1762. PMID 22505857
- [Background] Alberio T, Bossi AM, Milli A, Parma E, Gariboldi MB, Tosi G, Lopiano L, Fasano M. Proteomic analysis of dopamine and alpha-synuclein interplay in a cellular model of Parkinson's disease pathogenesis. FEBS J. 2010 Dec;277(23):4909-19. doi: 10.1111/j.1742-4658.2010.07896.x. Epub 2010 Oct 26. PMID 20977677
- [Background] Venda LL, Cragg SJ, Buchman VL, Wade-Martins R. alpha-Synuclein and dopamine at the crossroads of Parkinson's disease. Trends Neurosci. 2010 Dec;33(12):559-68. doi: 10.1016/j.tins.2010.09.004. Epub 2010 Oct 18. PMID 20961626
- [Background] Taylor TN, Potgieter D, Anwar S, Senior SL, Janezic S, Threlfell S, Ryan B, Parkkinen L, Deltheil T, Cioroch M, Livieratos A, Oliver PL, Jennings KA, Davies KE, Ansorge O, Bannerman DM, Cragg SJ, Wade-Martins R. Region-specific deficits in dopamine, but not norepinephrine, signaling in a novel A30P alpha-synuclein BAC transgenic mouse. Neurobiol Dis. 2014 Feb;62:193-207. doi: 10.1016/j.nbd.2013.10.005. Epub 2013 Oct 10. PMID 24121116